CLINICAL TRIAL: NCT03487068
Title: Assessment of Renal Changes in Patients With Non Alcoholic Fatty Liver Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Maiada Mohie Eldin Ibrahim, Resident Doctor Of Gastroenterology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Renal changes with NAFLD
Record Dates: First submitted 2018-03-22; First posted 2018-04-03 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-03

CONDITIONS: Non-Alcoholic Fatty Liver Disease; Chronic Kidney Diseases
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with NAFLD (Other)
  Interventions: Device: The FibroScan device

INTERVENTIONS:
Device: The FibroScan device — The Fibroscan device (Echosens) works by measuring shear wave velocity. In this technique, a 50-MHz wave is passed into the liver from a small transducer on the end of an ultrasound probe. The probe also has a transducer on the end that can measure the velocity of the shear wave (in meters per second) as this wave passes through the liver. The shear wave velocity can then be converted into liver stiffness, which is expressed in kilopascals. Essentially, the technology measures the velocity of the sound wave passing through the liver and then converts that measurement into a liver stiffness measurement; the entire process is often referred to as liver ultrasonographic elastography.

SUMMARY:
Assess the renal changes in patients with non-alcoholic fatty liver (NAFLD).

DETAILED DESCRIPTION:
* Non-alcoholic fatty liver disease (NAFLD) is the accumulation of fat (>5%) in liver cells in the absence of excessive alcohol intake or other causes of liver disease. The histologic spectrum of NAFLD ranges from simple steatosis to non-alcoholic steatohepatitis (NASH), liver fibrosis, and cirrhosis. This disease affects up to 30% of the general population in Western countries, especially in patients with metabolic syndrome, obesity, and type II diabetes.
* Accumulating epidemiologic evidence indicates that NAFLD not only affects the liver but also increases the risk of extra-hepatic diseases such as type 2 diabetes mellitus, metabolic syndrome, hypertension, cardiovascular or cerebrovascular diseases, and chronic kidney disease.
* Chronic kidney disease (CKD) is defined by decreased estimated glomerular filtration rate (eGFR) and/or the presence of significant proteinuria. Its prevalence is ~ 4.3 - 13% in general population, but it is expected to increase and ~ 50% of these patients develop end-stage renal disease. Recently, CKD is significantly higher in patients with NAFLD than patients without.
* Several studies have demonstrated that NAFLD independently contributes to increasing the risk of CKD where NAFLD and CKD may share many common cardio-metabolic risk factors e.g. insulin resistance, chronic inflammation, and obesity.
* The exact pathophysiologic mechanisms linking NAFLD to CKD are not completely understood, however, there is increased production of various proinflammatory cytokines, reactive oxygen species, TNF-α, C-reactive protein (CRP), and IL-6 by hepatocytes and non-parenchymal cells (Kupffer cells and hepatic stellate cells) that can link NAFLD and CKD. In addition, altered rennin-angiotensin system activation can be involved.
* Several western studies had evaluated the relationship between NAFLD and CKD and shown the prevalence of CKD in NAFLD patients between 4 - 40%.
* An analysis of the United Network Organ Sharing (UNOS) data base during the years (2002-2011) revealed that 35% of the patients transplanted for NAFLD-related cirrhosis progressed to stage 3-4 CKD within 2 years after liver transplantation in comparison to 10% of patients transplanted for other etiologies.
* Despite these findings CKDs often goes unrecognized and The Third National Health and Nutrition survey (NHANESIII), among all individuals with moderately decreased GFR (less than 60ml/min; stage 3) reported the awareness was approximately 8%.
* There is still very little prospective studies and data linking NAFLD to CKD, and it is lacking in the middle east region.

ELIGIBILITY:
Inclusion Criteria:

•Patients diagnosed as NAFLD by abdominal ultrasonography, Fibroscan, NAFLD fibrosis score and FIB-4 score

Exclusion Criteria:

* Patients with diabetes and/or hypertension.
* Patients with chronic renal disease.
* Patients with urinary tract infections.
* Patients on medications affecting the kidney (eg: NSAIDs,..etc)
* Patients with chronic liver disease other than NAFLD (chronic hepatitis; viral B,C, autoimmune etc).
* Alcohol consumption.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-30 (Estimated); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-05-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of renal changes in patients with non-alcoholic fatty liver disease | baseline
  Measuring renal changes especially glomerular and interstitial pathologies which will lead to chronic kidney disease in patients with non alcoholic fatty liver disease.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Castera L. Diagnosis of non-alcoholic fatty liver disease/non-alcoholic steatohepatitis: Non-invasive tests are enough. Liver Int. 2018 Feb;38 Suppl 1:67-70. doi: 10.1111/liv.13658. PMID 29427494
- [Background] Sinn DH, Kang D, Jang HR, Gu S, Cho SJ, Paik SW, Ryu S, Chang Y, Lazo M, Guallar E, Cho J, Gwak GY. Development of chronic kidney disease in patients with non-alcoholic fatty liver disease: A cohort study. J Hepatol. 2017 Dec;67(6):1274-1280. doi: 10.1016/j.jhep.2017.08.024. Epub 2017 Sep 20. PMID 28870674